CLINICAL TRIAL: NCT01223443
Title: Sealing Moderate Coronary Saphenous VEin Graft Lesions With Paclitaxel-Eluting Stents as a New Approach to MainTaining VeIn Graft Patency and Reducing Cardiac Events
Brief Title: Sealing Moderate Coronary Saphenous VEin Graft Lesions With Paclitaxel-Eluting Stents
Acronym: VELETI II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was prematurely stopped due to slow patient enrolment.
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Collaborators: Boston Scientific Corporation (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VELETI II
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Coronary Artery Bypass Grafting; Drug Eluting Stent; Saphenous Vein Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI-stenting (Experimental): Stenting the moderate SVG lesion with the paclitaxel stent
  Interventions: Device: Paclitaxel eluting stent
- Standard medical treatment (No Intervention)

INTERVENTIONS:
Device: Paclitaxel eluting stent — Patients are randomized to either stenting the moderate SVG lesion with the paclitaxel stent or standard medical treatment
  Arms: PCI-stenting

SUMMARY:
Hypothesis: Sealing moderate SVG lesions with paclitaxel-eluting stents reduces cardiac events (death, myocardial infarction, target vessel revascularization) over the duration of follow-up.

Primary objective: To evaluate the efficacy of stenting moderate SVG lesions with paclitaxel-eluting stents on reducing the first occurrence of the composite of cardiac death, myocardial infarction or repeat revascularization related to the target SVG over the duration of follow-up (minimun of 2-year follow-up.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized study assessing the efficacy of stenting moderate SVG lesions (30% to 60% by visual estimation) with paclitaxel-eluting stents in the prevention of SVG atherosclerosis progression and cardiac events at follow-up. Patients with previous coronary bypass surgery with SVG implantation undergoing coronary angiography by clinical indication will be screened. If the patient has a moderate lesion at any level of the SVGs it will be includable in the study. After inclusion, the patients will be randomized to either stenting the moderate SVG lesion with the taxus stent or standard medical treatment. Following this procedure, all patients will have follow-up visits by telephone or clinic at 30 days, 180 days, 1 year, and yearly until the common study end date. The duration of the study will be approximately 4 years with a minimun of 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for cardiac catheterization and SVG angiography
2. Presence of at least one SVG lesion of 30% to 60% diameter stenoses, by visual estimation, which is not the culprit lesion* responsible for the clinical syndrome of the patient

   *If the target lesion is located in the same SVG than the culprit lesion (if present) it has to be at least 4 cm far from the stented segment)
3. Written informed consent

Exclusion Criteria:

1. Patient < 18 years old
2. Ejection fraction < 30%
3. Renal insufficiency with creatinine > 200 μmol/l
4. Presence of more than 2 moderate SVG stenoses in a single SVG or significant diffuse SVG disease defined as disease covering more than half of the length of the SVG
5. Presence of more than 2 SVGs with moderate SVG stenoses
6. Unsuccessful angioplasty (residual stenosis >30% and/or TIMI flow <3) of any other lesion treated during the same procedure (culprit lesions will be treated before patient randomization)
7. Any significant complication occurring during the angioplasty of the culprit lesion(s) during the same procedure
8. SVG lesion located at the distal anastomosis
9. SVG lesions located at the proximal anastomosis (lesion length < 5 mm from the SVG ostium)
10. Lesion length >25 mm
11. SVGs ≤ 3 years ago
12. Cardiogenic shock
13. Remaining coronary or SVG lesion(s) with treatment (PCI or CABG) planned within the following year
14. Pregnancy
15. Contraindication to aspirin and/or thienopyridine/ticagrelor treatment
16. Allergy to paclitaxel
17. Any disease with a limiting life-expectancy (less than 2 years)
18. Need for chronic anticoagulation treatment
19. Definite presence or high suspicion of thrombus or ulceration in the target lesion
20. Target lesion located in the same SVG as the culprit lesion (if present) and distance between the target lesion and the most proximal or distal part of the stent implanted at the culprit lesion < 4 cm
21. Vein graft diameter < 2.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-04; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The first occurrence of the composite of cardiac death, myocardial infarction or coronary revascularization related to the target SVG over the duration of follow-up. | 60 months

SECONDARY OUTCOMES:
1-First occurrence of the composite of cardiac death, myocardial infarction or coronary revascularization over the duration of follow-up. | 60 months
2-Cardiac death and myocardial infarction; repeat revascularization; and hospitalization due to an acute coronary syndrome. | 60 months
3-Total medical costs (at index hospitalization and at follow-up). | 60 months
4-Costs per major adverse cardiac event (cardiac death, myocardial infarction, revascularization) prevented. | 60 months
5-Severe (>60%) SVG lesions or SVG occlusion at the target SVG at 2-year follow-up as determined by 3D computed-tomography. | 60 months
6-Major bleeding complications defined according to the REPLACE-II criteria over the duration of follow-up. | 60 months
7-Stent thrombosis defined and classified according to the Academic Research Consortium criteria. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes-Cabau, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Rodes-Cabau J, Jolly SS, Cairns J, Mansour S, L'Allier PL, Teefy PJ, Graham JJ, Le May MR, Cantor WJ, Wood D, Balasubramanian K, DeLarochelliere R, Dzavik V; VELETI II Investigators (Sealing Moderate Coronary Saphenous Vein Graft Lesions With Paclitaxel-Eluting Stents). Sealing Intermediate Nonobstructive Coronary Saphenous Vein Graft Lesions With Drug-Eluting Stents as a New Approach to Reducing Cardiac Events: A Randomized Controlled Trial. Circ Cardiovasc Interv. 2016 Nov;9(11):e004336. doi: 10.1161/CIRCINTERVENTIONS.116.004336. PMID 27815344